CLINICAL TRIAL: NCT06453421
Title: Pulmonary Rehabilitation in the Chronically Critically Ill Patient: Prospective Study About Clinical Characteristics and the Response to Rehabilitation in This Patient Population and Search for Potential Predictive Factors
Brief Title: Pulmonary Rehabilitation in the Chronically Critically Ill Patient
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: PCCinRR-SP2022
Record Dates: First submitted 2024-05-14; First posted 2024-06-11 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Rehabilitation; Chronic Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic critical ill patients: Evaluation both of the clinical and pathophysiological characteristics of a group of chronically critical ill patients admitted to a pulmonary rehabilitation center and of their response to rehabilitation treatment
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Enrolled patients are subjected to a personalized respiratory rehabilitation treatment aimed both at weaning from the tracheostomy tube and at functional recovery

SUMMARY:
The goal of this observational study is to learn about the population of chronically critical ill patients who refer to respiratory rehabilitation units.

The main questions it aims to answer are:

* what are the clinical and pathophysiological characteristics of the population of chronically critical ill patients who refer to respiratory rehabilitation units after hospital admission with the need for prolonged invasive mechanical ventilation via tracheostomy?
* what is the response of this patient population to respiratory rehabilitation treatment in terms of functional recovery, weaning from invasive mechanical ventilation, weaning from tracheostomy tube, mortality and return to home?
* are there any appreciable indices at admission and/or in the first period of hospitalization which may have a prognostic significance both on short-term objectives (weaning from invasive mechanical ventilation, weaning from the tracheostomy tube) and in the medium-long term (survival, state of health)?

Participants will be subjected to a rehabilitation and weaning program consisting of:

* physical therapy,
* speech therapy,
* nutritional assessment and therapy,
* in subjects on invasive mechanical ventilation at admission a program of weaning and, if needed, shift from invasive to Non-Invasive Ventilation will be performed.

DETAILED DESCRIPTION:
Observational, prospective, non-profit study. The first aim is to define the clinical and pathophysiological characteristics of the population of chronic critically ill patients who refer to respiratory rehabilitation units after hospital admission with the need for prolonged invasive mechanical ventilation via tracheostomy.

The second aim is to identify the following aspects: evaluating the response of this particular patient population to respiratory rehabilitation treatment (functional recovery, weaning from invasive mechanical ventilation, decannulation and home discharge), knowing the mortality of this patient population and evaluating the existence of appreciable indices at admission and/or in the first period of hospitalization which may have a prognostic significance both on short-term objectives (weaning from invasive mechanical ventilation, weaning from the tracheostomy tube) and in the medium-long term (survival, state of health). This last aspect could also be useful for the early identification of patients who could benefit from rehabilitation treatment more than others and therefore to optimize the resources at our disposal.

The present study involves the collection of data from chronically critical patients who will be referred to the Rehabilitation Pneumology Unit of the Don Gnocchi Foundation in Florence after hospitalization in intensive care for respiratory failure with the need for prolonged invasive mechanical ventilation.

The prospective analysis will have a total duration of 6 months.

The enrolled patients will follow the standard care path provided by the center and in this context they will carry out the rehabilitation treatment both within the department and in the dedicated respiratory gym.

The variables of interest will be extracted from the medical records at the time of entry (T0) to the department and at the time of discharge (T1).

It is expected to enroll 220 patients under ordinary hospitalization at the unit of Rehabilitative Pneumology of the Don Gnocchi Foundation of Florence.

The default sample size was set based on the recruiting capacity of the center involved in the project.

The data will be retrieved from the medical records of patients belonging to the department.

The folders will be viewed by the main investigator and his collaborators and the data of interest and the reports of the instrumental tests will be extracted.

Starting from the clinical and anamnestic evaluation upon admission to the department, patients who fall within the inclusion criteria will be identified.

The data will be entered anonymously into a computerized database, in which each subject will be associated with an alphanumeric identification code. The correspondence between the patients' name and numerical identity (progressive enrollment number) will be recorded in a separate table (association key) kept by the principal investigator.

The paper data relating to the study will be stored in an archive accessible only to the Principal Investigator, while the electronic data will be stored on servers located in the territory of the European Union on physical archives protected by double key encryption systems.

During the duration of the study, access to the computerized and anonymized database will be limited to the principal investigator, who may extend access to identified collaborators. The anonymized data will be retained for a period of 7 years after the conclusion of the study. Once the retention period indicated above has expired, the data will be made anonymous so that it is no longer possible to trace, directly or indirectly, the identity of the interested party. The anonymized data may be reused for subsequent research and therefore stored by the joint owners indefinitely.

For the analysis of the primary objective, a descriptive statistic will be used through which the clinical and clinical-functional variables recorded at admission (T0) will be presented. In particular, for continuous variables (or similar to such, e.g. age, Barthel score) mean and standard deviation or median and interquartile range will be used, depending on whether the variables have a normal distribution or not, as descriptors respectively of central tendency and dispersion. The normality or otherwise of the distribution of each variable will be verified by evaluating the asymmetry and kurtosis parameters of the distribution itself. As regards dichotomous variables (e.g. presence of infections), the frequency values in the observed sample and the relative percentages will be reported.

For the analysis of the first secondary objective, a comparison will be made between the values recorded at T0 and at discharge (T1) for the clinical and clinical-functional variables that require a reassessment at T1. The comparison will be carried out using a T-test for paired measures or a Wilcoxon Signed-Rank Test in the case of continuous variables, depending on whether or not they have an approximately normal distribution. In the case of categorical/ordinal variables, the Wilcoxon Signed-Rank Test will be used and the McNemar's test in the case of dichotomous variables. For all tests a p-value<0.05 will be considered significant.

For the analysis of the second and third secondary objectives, logistic regression models will be used to evaluate the association between the independent variables (variables recorded at admission and their changes in the first weeks) and the dependent variables (weaning from invasive mechanical ventilation, weaning from tracheostomy tube, survival and health status).

Furthermore, the changes in parameters measured at admission and at discharge will be compared through repeated measures analyses. In particular, for continuous variables, a repeated measures ANOVA test or a Friedman test will be used, depending on whether the variables have a normal distribution or not. For dichotomous variables, a Cochran's Q test will be used. For all tests, a p-value<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years;
* episode of acute or acute-on-chronic respiratory failure with the need for prolonged invasive mechanical ventilation via tracheostomy

Exclusion Criteria:

condition of clinical instability such as to make it necessary to transfer the patient to acute hospital within the first 7 days of hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory failure who have undergone prolonged invasive mechanical ventilation via tracheostomy.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-08-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients weaned from the tracheostomy tube | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  for each patient the presence of the tracheostomy tube and its possible removal are assessed
Number of patients weaned from invasive mechanical ventilation | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  for each patient the need for invasive mechanical ventilation and its possible removal are assessed
arterial blood gas analysis | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  evaluation of respiratory exchanges in terms mainly of oxygen blood pressure (mmHg) and of carbon dioxide blood pressure (mmHg).
functional independence measure (FIM) scale | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  An international standard for measuring disability, with a score from 18 to 126 where higher values correspond to a greater level of autonomy
Modified barthel index (mBI) | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  An ordinal scale used to measure a subject's performance in Activities of Daily Living (ADL), with a score from 0 to 100 where higher values correspond to a greater level of autonomy
Short Physical Performance Battery (SPPB) | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  A group of measures that combines the results of the gait speed, chair stand and balance tests. It can be useful as a predictive tool for possible disability and can aid in the monitoring of function. With a score from 0 to 12 where higher values correspond to a better motor function.
Short Form 12 (SF12) | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  A self-reported measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure, with a score from 12 to 47 where lower values correspond to a better quality of life.
Pain evaluation | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  Intensity of the pain is assessed through the visual analogue scale (VAS). A 10 cm long visual scale where the length corresponds directly to the pain
Barthel dyspnea | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  An ordinal scale used to measure a subject's level of dyspnea while performing Activities of Daily Living (ADL), with a score from 0 to 100 where lower values correspond to a greater level of dyspnea.
Hospital Anxiety and Depression Scale (HADS) | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  A self-reported measure, made up of 14 items, 7 for the evaluation of anxiety and 7 for depression. For both anxiety and depression the score ranges from 0 to 21. The higher scores correspond to a greater probability of being affected by the pathology.
Malnutrition Universal Screening Tool (MUST) scale | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  A screening tool to identify malnourished adults, at risk of malnutrition (undernutrition) or obesity. It has a score ranging from 0 to 6. The lower score corresponds to a lower risk of malnutrition.
Change in nutritional status from admission to discharge | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  Global Leadership Initiative on Malnutrition (GLIM) criteria are 5 diagnostic criteria to assess malnutrition that include 3 phenotypic (weight loss, low body mass index and reduced muscle mass) and 2 etiologic (reduced food intake/assimilation, and inflammation /disease burden) criteria. To diagnose malnutrition at least 1 phenotypic criterion and 1 etiologic criterion should be present.
Montreal Cognitive Assessment (MoCA) | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  The MoCA is a tool for rapid screening of mild cognitive impairment. It evaluates different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructive skills, abstraction, calculation and orientation. The maximum possible score is 30 points; an equal score or above 26 is considered normal.
Functional Oral Intake Scale (FOIS) | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  A tool to assess functional oral intake of food and liquids in patients with oropharyngeal dysphagia. The score ranges from 1 (no oral intake) to 7 (total oral intake with no restrictions).
Medical Research Council (MRC) Scale | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  The MRC Scale is a scale of 6 values, ranging from 0 to 5, for measuring strength through the observation of muscle movements and behavior for grades from 0 to 3, and the administration of manual muscle tests for grades 4 and 5. It consists of a strength attribution score, ranging from 0 (absence of contraction) to 5 (normal strength).
Modified Rankin Scale (MRS) | From date of randomization until the date of discharge or date of hospitalization or death from any cause, whichever came first, assessed up to 1 year .
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of patients. The scale runs from 0-6, running from perfect health without symptoms (0) to death (6).

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Chellini, MD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi ONLUS, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Garnacho-Montero J, Amaya-Villar R, Garcia-Garmendia JL, Madrazo-Osuna J, Ortiz-Leyba C. Effect of critical illness polyneuropathy on the withdrawal from mechanical ventilation and the length of stay in septic patients. Crit Care Med. 2005 Feb;33(2):349-54. doi: 10.1097/01.ccm.0000153521.41848.7e. PMID 15699838
- [Background] Laghi F, Cattapan SE, Jubran A, Parthasarathy S, Warshawsky P, Choi YS, Tobin MJ. Is weaning failure caused by low-frequency fatigue of the diaphragm? Am J Respir Crit Care Med. 2003 Jan 15;167(2):120-7. doi: 10.1164/rccm.200210-1246OC. Epub 2002 Oct 31. PMID 12411288
- [Background] Demoule A, Jung B, Prodanovic H, Molinari N, Chanques G, Coirault C, Matecki S, Duguet A, Similowski T, Jaber S. Diaphragm dysfunction on admission to the intensive care unit. Prevalence, risk factors, and prognostic impact-a prospective study. Am J Respir Crit Care Med. 2013 Jul 15;188(2):213-9. doi: 10.1164/rccm.201209-1668OC. PMID 23641946
- [Background] Jung B, Moury PH, Mahul M, de Jong A, Galia F, Prades A, Albaladejo P, Chanques G, Molinari N, Jaber S. Diaphragmatic dysfunction in patients with ICU-acquired weakness and its impact on extubation failure. Intensive Care Med. 2016 May;42(5):853-861. doi: 10.1007/s00134-015-4125-2. Epub 2015 Nov 16. PMID 26572511
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Background] Dres M, Dube BP, Mayaux J, Delemazure J, Reuter D, Brochard L, Similowski T, Demoule A. Coexistence and Impact of Limb Muscle and Diaphragm Weakness at Time of Liberation from Mechanical Ventilation in Medical Intensive Care Unit Patients. Am J Respir Crit Care Med. 2017 Jan 1;195(1):57-66. doi: 10.1164/rccm.201602-0367OC. PMID 27310484
- [Background] Epstein SK. Anatomy and physiology of tracheostomy. Respir Care. 2005 Apr;50(4):476-82. PMID 15807905
- [Background] Carson SS. Definitions and epidemiology of the chronically critically ill. Respir Care. 2012 Jun;57(6):848-56; discussion 856-8. doi: 10.4187/respcare.01736. PMID 22663962
- [Background] Carson SS, Bach PB. The epidemiology and costs of chronic critical illness. Crit Care Clin. 2002 Jul;18(3):461-76. doi: 10.1016/s0749-0704(02)00015-5. PMID 12140908
- [Background] Kahn JM, Benson NM, Appleby D, Carson SS, Iwashyna TJ. Long-term acute care hospital utilization after critical illness. JAMA. 2010 Jun 9;303(22):2253-9. doi: 10.1001/jama.2010.761. PMID 20530778
- [Background] Confalonieri M, Gorini M, Ambrosino N, Mollica C, Corrado A; Scientific Group on Respiratory Intensive Care of the Italian Association of Hospital Pneumonologists. Respiratory intensive care units in Italy: a national census and prospective cohort study. Thorax. 2001 May;56(5):373-8. doi: 10.1136/thorax.56.5.373. PMID 11312406
- [Background] Mifsud Bonnici D, Sanctuary T, Warren A, Murphy PB, Steier J, Marino P, Pattani H, Creagh-Brown BC, Hart N. Prospective observational cohort study of patients with weaning failure admitted to a specialist weaning, rehabilitation and home mechanical ventilation centre. BMJ Open. 2016 Mar 8;6(3):e010025. doi: 10.1136/bmjopen-2015-010025. PMID 26956162
- [Background] Hannan LM, Tan S, Hopkinson K, Marchingo E, Rautela L, Detering K, Berlowitz DJ, McDonald CF, Howard ME. Inpatient and long-term outcomes of individuals admitted for weaning from mechanical ventilation at a specialized ventilation weaning unit. Respirology. 2013 Jan;18(1):154-60. doi: 10.1111/j.1440-1843.2012.02266.x. PMID 22985330
- [Background] Schonhofer B, Euteneuer S, Nava S, Suchi S, Kohler D. Survival of mechanically ventilated patients admitted to a specialised weaning centre. Intensive Care Med. 2002 Jul;28(7):908-16. doi: 10.1007/s00134-002-1287-5. Epub 2002 Apr 24. PMID 12122529
- [Background] Dasgupta A, Rice R, Mascha E, Litaker D, Stoller JK. Four-year experience with a unit for long-term ventilation (respiratory special care unit) at the Cleveland Clinic Foundation. Chest. 1999 Aug;116(2):447-55. doi: 10.1378/chest.116.2.447. PMID 10453875
- [Background] Quinnell TG, Pilsworth S, Shneerson JM, Smith IE. Prolonged invasive ventilation following acute ventilatory failure in COPD: weaning results, survival, and the role of noninvasive ventilation. Chest. 2006 Jan;129(1):133-9. doi: 10.1378/chest.129.1.133. PMID 16424423
- [Background] Heinemann F, Budweiser S, Jorres RA, Arzt M, Rosch F, Kollert F, Pfeifer M. The role of non-invasive home mechanical ventilation in patients with chronic obstructive pulmonary disease requiring prolonged weaning. Respirology. 2011 Nov;16(8):1273-80. doi: 10.1111/j.1440-1843.2011.02054.x. PMID 21883681
- [Background] Rose L, Fraser IM. Patient characteristics and outcomes of a provincial prolonged-ventilation weaning centre: a retrospective cohort study. Can Respir J. 2012 May-Jun;19(3):216-20. doi: 10.1155/2012/358265. PMID 22679615
- [Background] Scheinhorn DJ, Hassenpflug MS, Votto JJ, Chao DC, Epstein SK, Doig GS, Knight EB, Petrak RA; Ventilation Outcomes Study Group. Post-ICU mechanical ventilation at 23 long-term care hospitals: a multicenter outcomes study. Chest. 2007 Jan;131(1):85-93. doi: 10.1378/chest.06-1081. PMID 17218560
- [Background] Stoller JK, Xu M, Mascha E, Rice R. Long-term outcomes for patients discharged from a long-term hospital-based weaning unit. Chest. 2003 Nov;124(5):1892-9. doi: 10.1378/chest.124.5.1892. PMID 14605065
- [Background] Pilcher DV, Bailey MJ, Treacher DF, Hamid S, Williams AJ, Davidson AC. Outcomes, cost and long term survival of patients referred to a regional weaning centre. Thorax. 2005 Mar;60(3):187-92. doi: 10.1136/thx.2004.026500. PMID 15741433
- [Background] Aboussouan LS, Lattin CD, Anne VV. Determinants of time-to-weaning in a specialized respiratory care unit. Chest. 2005 Nov;128(5):3117-26. doi: 10.1378/chest.128.5.3117. PMID 16304251
- [Background] Latriano B, McCauley P, Astiz ME, Greenbaum D, Rackow EC. Non-ICU care of hemodynamically stable mechanically ventilated patients. Chest. 1996 Jun;109(6):1591-6. doi: 10.1378/chest.109.6.1591. PMID 8769516
- [Background] Gracey DR, Hardy DC, Naessens JM, Silverstein MD, Hubmayr RD. The Mayo Ventilator-Dependent Rehabilitation Unit: a 5-year experience. Mayo Clin Proc. 1997 Jan;72(1):13-9. doi: 10.4065/72.1.13. PMID 9005279